CLINICAL TRIAL: NCT02184130
Title: Altered Vestibular Perception by Virtual Lesions of Cerebral and Cerebellar Structures Using Repetitive Transcranial Magnetic Stimulation - Implications for Human Vestibular Dysfunction
Brief Title: Altered Vestibular Perception and Transcranial Magnetic Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient funds and participants, thus terminated
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: tms_percept_zurich
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Verticality Perception; Self-motion Perception
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMS (Experimental)
  Interventions: Other: transcranial magnetic stimulation and motion stimuli

INTERVENTIONS:
Other: transcranial magnetic stimulation and motion stimuli

SUMMARY:
The long-term goal of this research is to advance our knowledge of how information from the labyrinth is brought to perception and how adaptation to vestibular imbalance influences motion sensation. Patients with vestibular disorders frequently have disabling disturbances of perception. Related to these symptoms is that large areas of the cerebral hemispheres and the cerebellum receive information from the vestibular, visual and somatosensory systems that is integrated within a vestibular cortical network into an accurate perception of spatial orientation. Interrupting the pathways that process information about the direction of gravity and angular velocity leads to impairment of the internal estimate of gravity and the perception of body motion. The strategy of this research is to use repetitive transcranial magnetic stimulation (rTMS) to produce transient focal lesions that allow study of acute loss of function within the central vestibular pathways at the very beginning of adaptation. Our underlying hypothesis is that the immediate effects of a lesion in the cerebellum will be to affect ocular motor control of vestibular reflexes and perception alike but with a cortical lesion there will be dissociation between ocular motor control and perception. This research helps to understand the mechanisms involved in the perception of vestibular information and the cerebellar influence on processing vestibular input and offers a unique opportunity to make major inroads into the understanding and eventually treatment of the often incapacitating symptoms of patients with vestibular disease

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-70
2. informed consent

Exclusion Criteria:

1. disturbed consciousness
2. other neurological or systemic disorder which can cause dementia or cognitive dysfunction
3. prior history of a major psychiatric disorder
4. history of definite stroke
5. focal lesion on MRI exam
6. use of anxiolytic, antidepressant, neuroleptic or sedative medication
7. has MRI contraindication such as pacemaker, implanted pumps, shrapnel, etc. (full MRI screening form will be filled out).
8. History of seizure or a family history of epilepsy;
9. increased intracranial pressure, such as after infarctions or trauma
10. pregnancy or possibility of being pregnant unless precluded by a negative pregnancy test
11. history of any significant head trauma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
changes in verticality perception and self-motion perception after TMS (transcranial magnetic stimulation) | within 30min after TMS

SECONDARY OUTCOMES:
vestibulo-ocular reflex after TMS (transcranial magnetic stimulation) | within 30min after TMS

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Straumann, Prof MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland